CLINICAL TRIAL: NCT01656785
Title: 68Ga-BNOTA-PRGD2 PET/CT in Evaluation of Angiogenesis Following Stroke
Brief Title: 68Ga-BNOTA-PRGD2 PET/CT in Evaluation of Stroke
Acronym: GRGDS
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCHNM004
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2014-11

CONDITIONS: Stroke
Keywords: stroke; cerebrovascular disease; angiogenesis imaging; 68Ga-BNOTA-PRGD2; PET/CT
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders | interventions — 68gallium-BNOTA-PRGD2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Brain 68Ga-BNOTA-PRGD2 (Experimental): We will perform brain 68Ga-BNOTA-PRGD2 PET/CT on stroke patients to determine its value.
  Interventions: Drug: 68Ga-BNOTA-PRGD2

INTERVENTIONS:
Drug: 68Ga-BNOTA-PRGD2 — Intravenous injection of one dosage of 111MBq 68Ga-BNOTA-PRGD2 solution. Tracer doses of 68Ga-BNOTA-PRGD2 will be used to image angiogenesis of cerebral infarction areas by Positron Emission Tomography / computed tomography (PET/CT)
  Other Names: 68Ga-p-SCN-Bn-NOTA-PEG3-RGD2

SUMMARY:
This is an open-label brain PET/CT (positron emission tomography/computed tomography) study to investigate the diagnostic performance of 68Ga-BNOTA-PRGD2 in evaluation of stroke patients in convalescence. A single dose of nearly 111 MBq 68Ga-BNOTA-PRGD2 ( ≤ 40 µg BNOTA-PRGD2) will be intravenously injected into the patients. Visual and semi-quantitative method will be used to assess the PET/CT images. Changes of 18F-FDG PET/CT, enhanced brain MRI or CT, and any adverse events will be collected from the patients.

DETAILED DESCRIPTION:
Integrin αvβ3 is an important member of this receptor family and expressed preferentially on regenerative vascular endothelial cells, but not or very low on the quiescent vessel cells and other normal cells. The αvβ3 integrin is a key mediator of angiogenesis and thus may be an important diagnostic and therapeutic target associated with cerebrovascular repair processes after stroke.

The tri-peptide sequence of arginine-glycine-aspartic acid (RGD) can specifically bind to the integrin αvβ3 receptor. Accordingly, a variety of radiolabeled RGD-based peptides have been developed for non-invasive imaging of integrin αvβ3 expression via positron emission tomography (PET) or single photon emission computed tomography (SPECT) to monitor the angiogenesis in clinical Oncology and Cardiology. In Neurology, angiogenesis imaging based on integrin αvβ3 receptor has not been found in clinical trials, but preclinical animal studies showed it had great potential for clinical translation. Recently, series of RGD dimeric peptides with PEG linkers have been studied. The new types of RGD peptides showed much higher in vitro integrin αvβ3 binding affinity than the single RGD tri-peptide sequence. As a representative, 68Ga-BNOTA-PRGD2 could be easily prepared and exhibited excellent in vivo behavior in animal models and also tumor or myocardial infarction patients. No adverse reactions are observed in animal models or patients to date.

For the further interests in clinical translation of 68Ga-BNOTA-PRGD2, an open-label brain PET/CT study was designed to investigate diagnostic performance of 68Ga-BNOTA-PRGD2 in stroke patients in convalescence. A single dose of nearly 111 MBq 68Ga-BNOTA-PRGD2 ( ≤ 40 µg BNOTA-PRGD2) will be intravenously injected into the patients. Visual and semiquantitative method will be used to assess the PET/CT images. Changes of brain 18F-FDG PET/CT, enhanced brain MRI or CT, and any adverse events will be collected from the patients.

ELIGIBILITY:
Inclusion Criteria:

stroke patients in convalescence:

* Males and females, ≥30 years old
* Confirmed cerebral infarction diagnosis
* With brain CT or MRI scans

Exclusion Criteria:

* Have cerebral tumors or other kinds of cerebral diseases
* Females planning to bear a child recently or with childbearing potential
* Renal function: serum creatinine >3.0 mg/dL (270 μM/L)
* Liver function: any hepatic enzyme level more than 5 times upper limit of normal.
* Known severe allergy or hypersensitivity to IV radiographic contrast.
* Patients not able to enter the bore of the PET/CT scanner.
* Inability to lie still for the entire imaging time because of cough, pain, etc.
* Inability to complete the needed examinations due to severe claustrophobia, radiation phobia, etc.
* Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the Investigator, may significantly interfere with study compliance.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-02; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Visual and semiquantitative assessment (Standardized Uptake Values = SUVs) of cerebral infarction region, SUV ratios (SUVinfarction/SUV contralateral) | 1 year
  Visual analysis will be performed by consensus reading by at least 3 experienced nuclear medicine physicians. The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake values (SUVs) of suspicious region in the stroke area and the SUV ratios (SUVinfarction/SUV contralateral) will be measured.

SECONDARY OUTCOMES:
Adverse events collection | 1 year
  Adverse events within 5 days after the injection and PET/CT scanning will be collected and assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, PhD, Principal Investigator — Department of Nuclear Medicine, Peking Union Medical College Hospital
Locations (1):
- Department of Nuclear Medicine, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China